CLINICAL TRIAL: NCT06955494
Title: The Effect of the "Empowerment Network for Auditory-Cognitive Training (ENACT) Program" on Auditory Perception and Function, Cognitive Function and Health-related Quality of Life of Persons Living With Mild Cognitive Impairment
Brief Title: ENACT Program on Auditory Perception and Function, Cognitive Function and Health-related Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENACT-Pilot
Record Dates: First submitted 2025-03-18; First posted 2025-05-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss; Cognitive Impairment, Mild
Keywords: cognitive impairment; hearing loss
MeSH Terms: conditions — Hearing Loss; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The ENACT Program is an overall 12-week training and comprises of three phases as follows:
  1. Goal-oriented health counseling phase (1st - 2nd week) - A nurse consultation will be conducted in the center with the aim to identify the participants' experience of living with the hearing and cognitive impairment.
  2. Peer-assisted group-based auditory-cognitive training phase (3rd-8th week) - This phase is led and conducted by the nurse with the focus to provide combined group-based auditory and cognitive training (group size = 6) with support from the trained peers.
  3. Family engaged active-communication training phase (9th - 12th week) - This phase is to empower the PLwMCI and their primary caregivers on active communication strategies in the presence of hearing loss.
  In the 2nd and 3rd phase, the nurse will continue to monitor the goal attainment of the PLwMCI and make additional health counseling and goal adjustment accordingly.
Who Masked: Outcomes Assessor
Masking Description: The pilot randomized controlled trial will be conducted in two elderly community centers of a non-government organization in Hong Kong. Participants will be randomized into intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENACT program (Experimental): The ENACT Program is an overall 12-week training and comprises of three phases as follows:
  1. Goal-oriented health counseling phase (1st - 2nd week) - A nurse consultation will be conducted in the center with the aim to identify the participants' experience of living with the hearing and cognitive impairment.
  2. Peer-assisted group-based auditory-cognitive training phase (3rd-8th week) - This phase is led and conducted by the nurse with the focus to provide combined group-based auditory and cognitive training (group size = 6) with support from the trained peers.
  3. Family engaged active-communication training phase (9th - 12th week) - This phase is to empower the PLwMCI and their primary caregivers on active communication strategies in the presence of hearing loss.
  In the 2nd and 3rd phase, the nurse will continue to monitor the goal attainment of the PLwMCI and make additional health counseling and goal adjustment accordingly.
  Interventions: Other: Empowerment Network for Auditory-Cognitive Training (ENACT) Program
- Usual care (Placebo Comparator): Usual care will be provided to the control group which mainly covers the social activities offered by the affiliated center. The participants are requested not to join any activities relating to cognitive training or auditory training before the post-test data collection.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Empowerment Network for Auditory-Cognitive Training (ENACT) Program — The ENACT Program is an overall 12-week training and comprises of three phases as follows: 1. Goal-oriented health counseling phase (1st - 2nd week) - A nurse consultation will be conducted in the center with the aim to identify the participants' experience of living with the hearing and cognitive impairment. 2. Peer-assisted group-based auditory-cognitive training phase (3rd-8th week) - This phase is led and conducted by the nurse with the focus to provide combined group-based auditory and cognitive training (group size = 6) with support from the trained peers. 3. Family engaged active-communication training phase (9th - 12th week) - This phase is to empower the PLwMCI and their primary caregivers on active communication strategies in the presence of hearing loss. In the 2nd and 3rd phase, the nurse will continue to monitor the goal attainment of the PLwMCI and make additional health counseling and goal adjustment accordingly.
  Arms: ENACT program
Other: Usual Care — Usual care will be provided to the control group which mainly covers the social activities offered by the affiliated center. The participants are requested not to join any activities relating to cognitive training or auditory training before the post-test data collection.
  Arms: Usual care

SUMMARY:
Although previous studies indicated that tackling hearing loss may have a secondary benefit in improving cognitive function and delaying the onset of dementia, a more integrated care approach to optimize both hearing and cognitive function may be needed for individuals who already developed cognitive decline. To address the dual care needs for PwMCI and hearing impairment, it may be possible to integrate auditory training into cognitive training, as both of them are activity-based and focus on increasing the attention and working memory of an individual to engage in the auditory communication process. Moreover, auditory instruction is one of the core mediums in delivering cognitive training activities. It is highly possible to integrate the auditory training curricular to the corresponding administration process. To tackle the enhanced support need of individuals with dual functional impairment to engage in an integrated training protocol, strategies including a goal-oriented approach and peer support can be integrated to optimize the empowerment network. Including family members in the training is also important, as the auditory-communication process in everyday life would take place in the social interactional context.

This is a pilot mixed-method pilot study comprising a randomized controlled trial and a post-trail qualitative interview. A total of 62 participants will be recruited from two community centers. The inclusion criteria include mild cognitive impairment according to Petersen's criteria; with at least one-side hearing impairment as defined by a score of 2- or 3-digit test greater than the norm value on the integrated Digit-in-Noise (iDIN test); has a smartphone to access the online training materials; not received formal cognitive and auditory training in the past 6 months. After the baseline outcome evaluation, they will be randomized to receive the 12-week ENACT program or the usual care control. The nurse-led ENACT program comprises three phases, including i) the goal-oriented health counselling phase, ii) the peer-assisted group-based auditory-cognitive training phase, and iii) the family-engaged active-communication training phase. The outcome evaluation on hearing function, perceived benefit of auditory training, cognitive function, and HRQoL will be assessed at baseline, in the 12th and 18th weeks. Qualitative interviews will be conducted

DETAILED DESCRIPTION:
Research evidence on tackling the dual cognitive and hearing impairment is very limited. Although previous studies indicated that tackling hearing loss may have a secondary benefit on improving cognitive function and delay the onset of dementia, a more integrated care approach to optimize both hearing and cognitive function may be needed for individuals who already developed cognitive decline. In fact, cognitive training is a standard evidence-based care to managing MCI. It is timely to explore how the management of hearing loss can be integrated to cognitive training to tackle the dual impairment. To address the dual care needs for PwMCI and hearing impairment, it may be possible to integrate auditory training to cognitive training, as both of them are activity-based and focusing on increasing the attention and working memory of an individual to engage in the auditory-communication process. Moreover, auditory instruction is one of the core mediums in delivering cognitive training activities. It is highly possible to integrate the auditory training curricular to the corresponding administration process. To tackle the enhanced support need of individuals with dual functional impairment to engage in an integrated training protocol, strategies including goal-oriented approach and peer support can be integrated to optimize the empowerment network. Including family members in the training is also important, as the auditory-communication process in everyday life would take place in the social interactional context.

The target population is the persons living with mild cognitive impairment (PLwMCI) who have hearing impairment. MCI is defined by a score of 19-26 out of the 30 on the Montreal Cognitive Assessment (education adjusted), the presence of subjective memory complaint and preserved daily activity function. [30] Hearing impairment is identified by the integrated Digit-In-Noise (DIN) test developed by the Co-I (L Wong) with the results of 2- or 3-digit results greater than the norm value to indicate hearing loss. Other inclusion criteria include: i) available of primary caregiver in the family, ii) have smart phone to receive online training materials, iii) not receive formal cognitive or auditory training in the past 6 months, iv) no other sensory impairment, and v) consent to participate.

The 12-week Empowerment Network on Auditory-Cognitive Training (ENACT) Program aims to offer combined auditory and cognitive training to the PLwMCI with hearing loss. A person-centered approach is used to not only engage the PLwMCI in combined auditory-cognitive training, but also to empower them and their significant others to maintain better communication, social interaction and social engagement in everyday life. Empowerment network refers to the use of collaborative and partnership approach between the nurse, family member and peer health coach to optimize and sustain the training effects of ENACT program. The ENACT Program comprises of three phases as follows:

Goal-oriented health counseling phase (1st - 2nd week) - A nurse consultation will be conducted in the center with the aim to identify the participants' experience of living with the hearing and cognitive impairment, particularly on how it affects their daily living, social engagement, coping and adaptation. Education on how such functional decline set up a vicious cycle of further impairment will be given to motivate self-directed goal setting. An agreeable action plan with consideration of the clients' preference and resource will be developed. On the followed week, the nurse will conduct a telephone visit to follow up the action plan implementation and give additional support if needed.

Peer-assisted group-based auditory-cognitive training phase (3rd-8th week) - This phase is led and conducted by the nurse with the focus to provide combined group-based auditory and cognitive training (group size = 6) with support from the trained peers. The content for the six sessions is developed according to the hierarchy of auditory skills proposed by Erher which comprises four level of increasing difficulty including sound awareness, sound discrimination, sound identification and sound comprehension. Activities proposed by the Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) on working memory training, attention bias motivation, and cognitive interpretive training are integrated in planning the auditory training activities to achieve the dual benefit.[33] To better secure the participants' confidence and motivation in learning, the training will be commenced with low difficulty level with lower level auditory training, and progressively to incorporate more cognitive training activities and higher level auditory training. A total of 2-3 trained peer health coach will join the group session to facilitate the practice. Home exercise in format of audio-scripts and online response grid are developed, so that the health coach can better engage the participants via their preferred social platform such as WhatsApp's or WeChat for two times before the next group session. Each qualified health coach has received 12- hour training which covers effective communication with persons with auditory-cognitive impairment, instructions to administer auditory and cognitive training activities, and motivational strategies for older adults.

Family engaged active-communication training phase (9th - 12th week) - This phase is to empower the PLwMCI and their primary caregivers on active communication strategies in the presence of hearing loss. The content is developed according to Active Communication Education (ACE Program) which developed for adults with hearing loss. This phase will comprise 2 bi-weekly training sessions for the PLwMCI and 2 online training sessions with the involvement of the primary family caregivers. The online session is needed as effective communication take places in interactional and interpersonal context. The importance and strategies for the family to engage the PLwMCI in everyday decision-making and activity will also be highlighted.

In the 2nd and 3rd phase, the nurse will continue to monitor the goal attainment of the PLwMCI and make additional health counseling and goal adjustment accordingly.

This is a pilot mixed method study, comprising a randomized controlled trial and a post-trail qualitative interview. A total of 62 participants will be recruited from two community center. The inclusion criteria include mild cognitive impairment accordingly to the Petersen's criteria; with at least one-side hearing impairment as defined by a score of 2- or 3- digit test greater than the norm value on the integrated Digit-in-Noise (iDIN test); has a smartphone to access the online training materials; not received formal cognitive and auditory training in the past 6 months. After the baseline outcome evaluation, they will be randomized to receive the 12-week ENACT program or the usual care control. The nurse-led ENACT program comprises three phases including i) goal-oriented health counseling phase, ii) the peer-assisted group-based auditory-cognitive training phase, and iii) the family engaged active-communication training phase. The outcome evaluation on hearing function, perceived benefit of auditory training, the cognitive function and HRQoL will be assessed at baseline, 12th and 18th week. Qualitative interview with the PLwMCI, their family members and the peer health coach will be conducted to solicit their experience in the process.

The nurse will assess the baseline outcomes of the participants with the following validated measures before randomization. Another RA who has no information about the group assignment will conduct the post-test measure at the 12th and 18th week after the commencement of the intervention.

1. A battery of cognitive assessment will be used to evaluate various domains of cognition of the PLwMCI, including the Cantonese version of the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) for global cognition, the digit span-forward and backward test for attention and working memory, and Trail-Making Test Part A and B for complex attention, executive function and task switching. Multiple assessments are essential for detecting subtle cognitive changes.
2. The Glasgow Hearing Aid Benefit Profile will assess the self-perceived benefit of auditory training.
3. The Revised Hearing Handicap Inventory for the Elderly [37] to assess the perceived hearing loss.
4. The Short-From 12 Survey to measure the overall HRQoL as well as the physical and mental health.

Upon the completion of the ENACT Program, interviews will be conducted to the participants and their family caregivers in a dyadic format. Focus group interview will be conducted to health coach. The interviews will be audiotaped with the consent of the participants. Interview guides with open-ended questions are used to guide the interviews.

Data will be analyzed on an intention-to-treat basis. Skewed variables will be transformed before subjected to analyses. Baseline characteristics between the two arms of participants will be compared using t test, chi-square test or Fisher's exact test, as appropriate. Generalized Estimating Equation will be used to compare the differential changes on the health outcomes of the PLwMCI and family caregivers across the baseline, 12th week (T2) and 18th Week (T3) between the two study arms, with adjustment for a set of priori control variables including age, sex, educational level and other comorbidity burden. The findings will provide important insights on the feasibility, clients' perception and preliminary effect of an innovative care approach to tackle dual functional loss in PLwMCI with hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment accordingly to the Petersen's criteria
* With at least one-side hearing impairment as defined by a score of 2- or 3- digit test greater than the norm value on the integrated Digit-in-Noise (iDIN test)
* Has a smartphone to access the online training materials
* Not received formal cognitive and auditory training in the past 6 months.
* Available of primary caregiver in the family
* give consent to participate

Exclusion Criteria:

* moderate and severe cognitive impairment
* Other sensory impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons living with mild cognitive impairment (PLwMCI) who have hearing impairment
Enrollment: 62 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog) | Baseline (T0)
  Evaluate the cognitive domain function of the patient with dementia (PwD), scale from 0-70, with higher score indicating poor cognitive function.
Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog) | 12th week (T1) after baseline
  Evaluate the cognitive domain function of the patient with dementia (PwD), scale from 0-70, with higher score indicating poor cognitive function.
Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog) | 18th week (T2) after baseline
  Evaluate the cognitive domain function of the patient with dementia (PwD), scale from 0-70, with higher score indicating poor cognitive function.
The digit span-forward and backward test | Baseline (T0)
  Evaluate the attention and working memory of the patient with dementia, scales from 10 to 56, with higher score indicating better attention and working memory function
The digit span-forward and backward test | 12th week (T1) after baseline
  Evaluate the attention and working memory of the patient with dementia, scales from 10 to 56, with higher score indicating better attention and working memory function
The digit span-forward and backward test | 18th week (T2) after baseline
  Evaluate the attention and working memory of the patient with dementia, scales from 10 to 56, with higher score indicating better attention and working memory function
Trail-Making Test Part A and B | Baseline (T0)
  Evaluate the complex attention, executive function and task switching, with shorter time required to complete the task indicating better complex attention, executive function and task switching function
Trail-Making Test Part A and B | 12th week (T1) after baseline
  Evaluate the complex attention, executive function and task switching, with shorter time required to complete the task indicating better complex attention, executive function and task switching function
Trail-Making Test Part A and B | 18th week (T2) after baseline
  Evaluate the complex attention, executive function and task switching, with shorter time required to complete the task indicating better complex attention, executive function and task switching function

SECONDARY OUTCOMES:
Glasgow Hearing Aid Benefit Profile | Baseline (T0)
  Assess the self-perceived benefit of auditory training
Glasgow Hearing Aid Benefit Profile | 12th week (T1) after baseline
  Assess the self-perceived benefit of auditory training
Glasgow Hearing Aid Benefit Profile | 18th week (T2) after baseline
  Assess the self-perceived benefit of auditory training
Revised Hearing Handicap Inventory for the Elderly | Baseline (T0)
  Assess the perceived hearing loss, higher score means greater handicapping effect of a hearing impairment
Revised Hearing Handicap Inventory for the Elderly | 12th week (T1) after baseline
  Assess the perceived hearing loss, higher score means greater handicapping effect of a hearing impairment
Revised Hearing Handicap Inventory for the Elderly | 18th week (T2) after baseline
  Assess the perceived hearing loss, higher score means greater handicapping effect of a hearing impairment
12-Item Short-Form Health Survey | Baseline (T0)
  Measure the overall Health-Related Quality of Life as well as the physical and mental health, scale from 0-100, higher score indicates better quality of life
12-Item Short-Form Health Survey | 12th week (T1) after baseline
  Measure the overall Health-Related Quality of Life as well as the physical and mental health, scale from 0-100, higher score indicates better quality of life
12-Item Short-Form Health Survey | 18th week (T2) after baseline
  Measure the overall Health-Related Quality of Life as well as the physical and mental health, scale from 0-100, higher score indicates better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: SAU FUNG DORIS YU, PhD, Principal Investigator — HKU School of Nursing
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Petersen RC. Mild cognitive impairment as a diagnostic entity. J Intern Med. 2004 Sep;256(3):183-94. doi: 10.1111/j.1365-2796.2004.01388.x. PMID 15324362
- [Background] Laplante-Levesque A, Hickson L, Worrall L. Rehabilitation of older adults with hearing impairment: a critical review. J Aging Health. 2010 Mar;22(2):143-53. doi: 10.1177/0898264309352731. Epub 2010 Jan 7. PMID 20056812
- [Background] Hallberg LR, Hallberg U, Kramer SE. Self-reported hearing difficulties, communication strategies and psychological general well-being (quality of life) in patients with acquired hearing impairment. Disabil Rehabil. 2008;30(3):203-12. doi: 10.1080/09638280701228073. PMID 17852289
- [Background] Sprinzl GM, Riechelmann H. Current trends in treating hearing loss in elderly people: a review of the technology and treatment options - a mini-review. Gerontology. 2010;56(3):351-8. doi: 10.1159/000275062. Epub 2010 Jan 12. PMID 20090297
- [Background] Jorgensen LE, Messersmith JJ. Impact of Aging and Cognition on Hearing Assistive Technology Use. Semin Hear. 2015 Aug;36(3):162-74. doi: 10.1055/s-0035-1555119. PMID 27516716
- [Background] Gallagher NE, Woodside JV. Factors Affecting Hearing Aid Adoption and Use: A Qualitative Study. J Am Acad Audiol. 2018 Apr;29(4):300-312. doi: 10.3766/jaaa.16148. PMID 29664724
- [Background] Zheng H, Wong LLN, Hickson L. Barriers to hearing aid adoption among older adults in mainland China. Int J Audiol. 2023 Sep;62(9):814-825. doi: 10.1080/14992027.2022.2105263. Epub 2022 Aug 23. PMID 35997572
- [Background] Bucholc M, Bauermeister S, Kaur D, McClean PL, Todd S. The impact of hearing impairment and hearing aid use on progression to mild cognitive impairment in cognitively healthy adults: An observational cohort study. Alzheimers Dement (N Y). 2022 Feb 22;8(1):e12248. doi: 10.1002/trc2.12248. eCollection 2022. PMID 35229022
- [Background] Dawes P, Wolski L, Himmelsbach I, Regan J, Leroi I. Interventions for hearing and vision impairment to improve outcomes for people with dementia: a scoping review. Int Psychogeriatr. 2019 Feb;31(2):203-221. doi: 10.1017/S1041610218000728. Epub 2018 Sep 24. PMID 30244688
- [Background] Chen L, Zhou R. Does self-reported hearing difficulty decrease older adults' cognitive and physical functioning? The mediating role of social isolation. Maturitas. 2020 Nov;141:53-58. doi: 10.1016/j.maturitas.2020.06.011. Epub 2020 Jun 20. PMID 33036703
- [Background] Mitchell AJ, Shiri-Feshki M. Rate of progression of mild cognitive impairment to dementia--meta-analysis of 41 robust inception cohort studies. Acta Psychiatr Scand. 2009 Apr;119(4):252-65. doi: 10.1111/j.1600-0447.2008.01326.x. Epub 2008 Feb 18. PMID 19236314
- [Background] Lawrence BJ, Jayakody DMP, Bennett RJ, Eikelboom RH, Gasson N, Friedland PL. Hearing Loss and Depression in Older Adults: A Systematic Review and Meta-analysis. Gerontologist. 2020 Apr 2;60(3):e137-e154. doi: 10.1093/geront/gnz009. PMID 30835787
- [Background] Dalton DS, Cruickshanks KJ, Klein BE, Klein R, Wiley TL, Nondahl DM. The impact of hearing loss on quality of life in older adults. Gerontologist. 2003 Oct;43(5):661-8. doi: 10.1093/geront/43.5.661. PMID 14570962
- [Result] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT06955494/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT06955494/ICF_001.pdf